CLINICAL TRIAL: NCT03575221
Title: A Natural History of the Collagen-Related Disorder Osteogenesis Imperfecta and the Genotype-Phenotype Correlation
Brief Title: Natural History of the Collagen-Related Disorder Osteogenesis Imperfecta and Genotype Phenotype Correlation
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180120; 18-CH-0120
Record Dates: First submitted 2018-06-28; First posted 2018-07-02 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10-07

CONDITIONS: Osteogenesis Imperfecta; Short Stature
Keywords: Osteogenesis Imperfecta; Collagen; Short Stature; Natural History
MeSH Terms: conditions — Osteogenesis Imperfecta; Dwarfism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrollees: Individuals with Osteogenesis Imperfecta

SUMMARY:
Background:

Osteogenesis Imperfecta (OI) is a connective tissue disorder. OI affects many aspects of a person s health and growth. It can cause frequent fractures, short stature, and bowing of the long bones. There is no known cure for OI so researchers want to learn more about it.

Objectives:

To obtain a natural history of the course of OI. To find changes in genes that affect the disease.

Eligibility:

People from birth to age 12 years with certain types of OI

People who previously had childhood data collected in certain other protocols

Design:

Participants will stay in the clinic for a few days each visit. Visits will be about every 3-4 months to age 5 then about every 6-12 months. Visits may include:

Medical history

Physical exam

Hearing test

Dental exam

Blood, urine, and heart tests

Breathing measured while wearing a clear plastic hood for about 30 minutes

Tests of motion, strength, and motor skills

X-rays of the left hand, chest, legs, and spine

Bone density scan. Participants will lie on a flat table while a very small dose of x-rays is passed through the body.

Computed tomography and magnetic resonance imaging scans. Participants will lie on an exam table that moves in and out a scanner.

Breathing tests using stickers on the chest, a light probe on a finger or foot, and a face mask

Ultrasound of the kidneys, ureters, and bladder

Questionnaires

A small section of skin removed from the arm or thigh

For some tests, participants may take medicine to make them sleepy.

Participants may give separate consent for photos to be taken.

DETAILED DESCRIPTION:
study Description:

This is a longitudinal study of the natural history of the collagen-related disorder osteogenesis imperfecta (OI), that includes enrolling new patients under the age of 12 years, along with an extended data collection from adult patients on whom previous childhood data was collected at the NIH.

Objectives:

Primary Objectives: 1) Identify and monitor longitudinal functional outcomes of individuals with collagen and collagen-related disorders, with focuses on identifying underlying contributing factors and comorbidities for scoliosis; gaining insight into occurrence and progression of cardiac valvular abnormalities; pathogenesis of primary lung parenchymal defects; and establish novel data relating to metabolism in OI and its relationship to obesity. 2) Correlate genotypic and phenotypic expression. 3) Identify genetic factors that modify the severity of clinical expression

Secondary Objectives: Adapt and develop standard of care management guidelines for individuals with collagen and collagen-related disorders.

Endpoints:

Primary Endpoints: 1) Clinical course, underlying pathogenesis, and comorbidities in the assessed systems in individuals with OI including for each focus: scoliosis progression across age, scoliosis progression relating to predictive factor, and scoliosis progression relating to mutation spectrum; time to development of valvular abnormality; development of pulmonary tissue abnormalities, presence/absence of pulmonary tissue abnormality, and time to development of pulmonary tissue abnormality; time to development of metabolic abnormality. 2) Correlation of phenotype relating to genotype. 3) Causes of morbidities in individuals with OI.

Secondary endpoints: Tolerability and feasibility of each measure of the clinical battery of assessments based on clinical observation.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet either #1 OR #2 of the following criteria:

1. Individuals previously enrolled in 97-CH-0064, or other NIH OI study protocols for whom childhood data were collected at the NIH.

   OR
2. Individuals from birth to age 12 years at enrollment to this protocol 18-CH-0120 with

a diagnosis of any of OI type III - XVIII or potential additional types.

Diagnosis of OI determined by identification of:

1. A mutation in one allele of genes causing autosomal dominant OI types

   (COL1A1, COL1A2, or IFITM5), OR
2. at least one mutation in genes that are indicative of the autosomal recessive OI types.

OR

Individuals with a clinical diagnosis of OI, and a mutation in one of the above genes identified through the Rare Bone disease screening protocol (04-CH-0077).

EXCLUSION CRITERIA:

* Individuals with the diagnosis of OI Type I.
* Individuals who cannot travel to the NIH because of their medical condition.
* Individuals who, in the opinion of the Investigator, are unable to comply with the protocol or have medical conditions that would potentially increase the risk of participation.

<TAB>

There are no exclusionary criteria related to race or gender for this protocol.

Ages: 1 Day to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals of all ages, races, genders, and nationalities@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Clinical course, underlying pathogenesis, and comorbidities in the assessed systems in individuals with OI | Ongoing
  clinical course
Correlation of genotype and phenotype | Ongoing
  genotype-phenotype correlations
Causes of morbidities in individuals with OI | Ongoing
  clinical course

SECONDARY OUTCOMES:
Tolerability and feasibility of each measure of the clinical battery of assessments based on clinical observation | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Joshua J Zimmerberg, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Once primary and secondary endpoints are met to be able to publish/share, we will create a plan to address the IPD sharing as well.

REFERENCES:
- [Derived] Gochuico BR, Hossain M, Talvacchio SK, Zuo MXG, Barton M, Dang Do AN, Marini JC. Pulmonary function and structure abnormalities in children and young adults with osteogenesis imperfecta point to intrinsic and extrinsic lung abnormalities. J Med Genet. 2023 Nov;60(11):1067-1075. doi: 10.1136/jmg-2022-109009. Epub 2023 May 16. PMID 37197785
- [Derived] Ballenger KL, Tugarinov N, Talvacchio SK, Knue MM, Dang Do AN, Ahlman MA, Reynolds JC, Yanovski JA, Marini JC. Osteogenesis Imperfecta: The Impact of Genotype and Clinical Phenotype on Adiposity and Resting Energy Expenditure. J Clin Endocrinol Metab. 2022 Jan 1;107(1):67-76. doi: 10.1210/clinem/dgab679. PMID 34519823
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-CH-0120.html